CLINICAL TRIAL: NCT01615159
Title: Maintenance of Recommended Sodium Intake
Acronym: SPICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JHSPH4135
Record Dates: First submitted 2012-04-16; First posted 2012-06-08 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2014-09

CONDITIONS: Maintenance of Recommended Sodium Intake
Keywords: Sodium; Diet; Urinary sodium excretion; Feeding study; Diet maintenance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self directed control (No Intervention)
- Behavior and lifestyle counseling (Active Comparator)
  Interventions: Behavioral: Behavior and lifestyle counseling

INTERVENTIONS:
Behavioral: Behavior and lifestyle counseling — 20 week intervention period where one group gets behavior and lifestyle counseling and the other group gets no active intervention
  Arms: Behavior and lifestyle counseling

SUMMARY:
The overall objective of this study is to assist the general public in achieving and maintaining the currently recommended sodium intake of 1500 mg/day through a reduced sodium intervention that emphasizes spices and herbs. The investigators hypothesize that after four weeks of eating a controlled diet, individuals will acclimate and adhere to a reduced sodium intake of 1500 mg/day and their taste preferences will change. The investigators also hypothesize that individuals in a low sodium behavioral intervention will maintain greater adherence to a dietary sodium intake of ≤ 1500 mg/day than individuals in a self-directed control group.

ELIGIBILITY:
Inclusion Criteria:

* Adults to whom the U.S. Dietary Guideline of < 1500 mg/day of sodium applies

Exclusion Criteria:

* Individuals with chronic kidney disease,
* Chronic poor health state,
* Pregnancy,
* Inability to complete feeding study,
* Investigator discretion

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urinary sodium excretion | Weeks 4, 24

SECONDARY OUTCOMES:
Change from baseline in preferences for level of sodium in food products | Weeks 4, 24
Percentage of people below 2300 mg/day sodium intake | Weeks 4, 24
Percentage of people below 1500 mg/day sodium intake | weeks 4, 24

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Anderson, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Anderson CA, Cobb LK, Miller ER 3rd, Woodward M, Hottenstein A, Chang AR, Mongraw-Chaffin M, White K, Charleston J, Tanaka T, Thomas L, Appel LJ. Effects of a behavioral intervention that emphasizes spices and herbs on adherence to recommended sodium intake: results of the SPICE randomized clinical trial. Am J Clin Nutr. 2015 Sep;102(3):671-9. doi: 10.3945/ajcn.114.100750. Epub 2015 Aug 12. PMID 26269371